CLINICAL TRIAL: NCT04384055
Title: Predicting Outcomes for Covid-19 Using Sonography
Acronym: POCUS
Status: Completed | Type: Observational
Sponsor: Stanford University (Other)
Responsible Party: Sponsor
Other Study IDs: IRB-55621
Record Dates: First submitted 2020-05-08; First posted 2020-05-12 (Actual); Last update posted 2021-12-03 (Actual); Status verified 2021-12

CONDITIONS: COVID-19; Pneumonia, Viral
MeSH Terms: conditions — COVID-19; Pneumonia, Viral

STUDY DESIGN:
Observational Model: Case-Control | Time Perspective: Prospective
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

GROUPS / COHORTS (2):
- Covid-19 Positive Patients: This group includes individuals who were diagnosed with Covid-19 based on reverse transcriptase polymerase chain reaction (RT-PCR) of the nasopharynx
  Interventions: Diagnostic Test: Lung Ultrasound
- Covid-19 Negative Patients: This group includes individuals who did NOT have a positive test for Covid-19 based on reverse transcriptase polymerase chain reaction (RT-PCR) of the nasopharynx.
  Interventions: Diagnostic Test: Lung Ultrasound

INTERVENTIONS:
Diagnostic Test: Lung Ultrasound — Lung ultrasound will be performed on patients undergoing investigation for covid-19 based on a nasopharyngeal PCR.

SUMMARY:
This study seeks to investigate the role of lung ultrasound in caring for Covid-19 positive patients and whether it can be used to predict patient deterioration. This information will be vital for healthcare workers who seek to identify Covid-19 pneumonia or patients at risk for deterioration early in the disease course.

DETAILED DESCRIPTION:
As Covid-19 continues to stress hospital-based resources (including personal protective equipment, ancillary staff availability, and imaging study utilization), it is important to assess whether alternative methods for evaluating patients can be utilized to appropriately triage and care for Covid-positive patients. Current limitations of caring for patients with Covid-19 include the exposure of ancillary healthcare workers (including radiological technicians) and the time/resources required to decontaminate traditional radiological equipment such as x-ray or computerized tomography (CT) machines.

Point-of-care ultrasound (POCUS) has the potential to transform healthcare delivery due to its diagnostic and therapeutic expediency. It can be quickly performed at the bedside by experienced clinicians. It it has been shown to reliably and accurately diagnose patients with a variety of lung diseases, including pneumonia. This study seeks to investigate the role of lung ultrasound in caring for Covid-19 positive patients and whether it can be used to predict patient deterioration. This information will be vital for healthcare workers who seek to identify the virus or patients at risk for deterioration early in the disease course. Moreover, it has the potential to reduce the need for x-rays or CTs for Covid-19 patients, which has the potential to alleviate a significant burden currently being placed on the healthcare system.

ELIGIBILITY:
Inclusion Criteria:

* Any adult (18 or more years of age) presenting to the emergency department with symptoms suspicious for Covid-19
* This individual underwent evaluation for Covid-19 via a nasopharyngeal RT-PCR
* This individual received a lung ultrasound by the study authors within 28 days from initial evaluation

Exclusion Criteria:

* Any individual who did not receive a lung ultrasound within 28 days from initial evaluation for covid-19 related illness

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: This population will include all persons under investigation (PUIs) for covid-19 presenting to the Stanford emergency department.
Sampling Method: Non-Probability Sample
Enrollment: 165 (Actual)
Dates: Start 2020-03-21 (Actual); Primary Completion 2021-11-15 (Actual); Study Completion 2021-11-15 (Actual)

PRIMARY OUTCOMES:
Number of Patients Experiencing Death, ICU Admission, Mechanical Ventilation, or Use of High-Flow Nasal Cannula | 28 days from initial evaluation
  Composite primary outcome of death, ICU admission, mechanical ventilation, or use of high-flow nasal cannula (categorical)

SECONDARY OUTCOMES:
Number of Patients Requiring Mechanical Ventilation | 28 days from initial evaluation
Number of Patients Requiring Supplemental Oxygen Usage | 28 days from initial evaluation
Duration of Supplemental Oxygen Usage | 28 days from initial evaluation
Length of Stay | 28 days from initial evaluation
  Duration of Hospitalization (days)
Characterization of Ultrasound Findings | 28 days from initial evaluation
  Descriptive analysis of ultrasound findings in Covid-19

CONTACTS AND LOCATIONS:
Overall Officials: Andre D Kumar, MD, MEd, Principal Investigator — Stanford University; Sally Graglia, MD, MPH, Principal Investigator — University of California, San Francisco
Locations (2):
- United States (2):
  - University of California San Francisco, San Francisco, California
  - Stanford University, Stanford, California

IPD SHARING:
Plan to Share IPD: No